CLINICAL TRIAL: NCT05485441
Title: The Community Nurse as a Public Health Determinant: a Quasi-experimental and Interventional Study of Promotion of Papillomavirus Vaccination in the School Population
Brief Title: The Community Nurse as a Public Health Determinant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Pasquale Stefanizzi, Assistant Professor, University of Bari Aldo Moro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UNIBA-HPV-001
Record Dates: First submitted 2022-07-12; First posted 2022-08-03 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: HPV; Nurse's Role

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Students (Experimental): The students
  Interventions: Other: Digital Educational Intervention
- Parents (Experimental): The parents
  Interventions: Other: Digital Educational Intervention

INTERVENTIONS:
Other: Digital Educational Intervention — The educational intervention will be provided (at T1) in two ways:
  (I) a video lecture in e-learning mode lasting about an hour, aimed at adolescents, using the School Institute's platform for distance education (II) the promotion of 2-minute "videopills" on the social channels most frequently used by students (dedicated youtube channel/school portal)

SUMMARY:
To date, there have been no interventional studies aimed at increasing HPV vaccination rates by making use of digital and involving all stakeholders within this process: nurses, physicians, caregivers, parents, and children/adolescents according to the PPI principle.

The primary objective of the project is to identify the effectiveness of a digital educational intervention, conducted by a multidisciplinary healthcare team and targeting adolescents of both sexes in secondary schools. The outcome measures will be: engagement, increased knowledge and self-efficacy, and vaccination uptake.

This project will identify new models for addressing public health needs. The secondary aim is to evaluate parents' attitudes toward vaccination pre- and post-intervention education.

A quasi-experimental, pre-post educational intervention study will be conducted by adopting a convenience sampling will be adopted at secondary schools in Bari (Puglia, Italy).

DETAILED DESCRIPTION:
The study will be carried out in a multiphasic mode. All steps are described below.

* First Phase (T0): the Community Nurses (CN) will send, via e-mail to all parents, a questionnaire aimed at investigating their children's vaccination status, hesitation to vaccination, sources of information, and information needs about vaccination. Then, upon prior arrangement with the school Principal, the CN will, in-person, distribute a questionnaire to all participating students to explore adolescents' knowledge about HPV vaccination, their involvement in vaccine decision-making, their feelings, and perceived self-efficacy.
* Second Phase (T1): the CN, after analyzing all the responses from the questionnaires administered to both parents (to investigate hesitations to vaccination) and students (on students' knowledge, involvement, feelings, self-efficacy), will set up an educational intervention, involving the members of expert (nurses and physicians' experts in public health).

Description of the educational intervention

The educational intervention will be provided (at T1) in two ways:

(I) a video lecture in e-learning mode lasting about an hour, aimed at adolescents, using the School Institute's platform for distance education, using audiovisual systems and slide presentations in Power Point format; learner-learner interactions will be possible through e-mail messages, real-time individual chats and asynchronous discussion forum conversations including comment sections.. The event will be recorded so that both adolescents and parents can access it at their convenience.

The educational content will generally take into account the following topic areas: a) basic information on HPV, modes of prevention and contagion, vaccination and sexual health; b) epidemiology on cervical cancer, incidence and mortality rates; c) preventive measures (vaccines, condoms, screening tests); and d) discussion with privileged witnesses who have experienced contagion.

No form of clinical counseling will be carried out during the video lectures. (II) the promotion of 2-minute "videopills" on the social channels most frequently used by students (dedicated youtube channel/school portal) in which clinical experts (pediatrician, hygienist, health care assistant, and CN) will raise awareness of the importance of HPV vaccination in adolescents, providing brief information on modes of transmission, prevention, and health effects of the virus.

- Third Phase (T2) - follow up In the last phase (three months after the intervention), parents will be contacted again by the CN, by telephone, to assess whether they have been vaccinated against HPV. At the same time, the effectiveness of the educational intervention will be evaluated by administering the same instruments used at T0.

ELIGIBILITY:
Inclusion Criteria:

* Students aged 11- 13 years and their parents.
* Students with disabilities, with visual and hearing impairment, with the suppor of their support teacher.

Exclusion Criteria:

* Students and/or parents who do not agree to participate
* Students and/or parents who do not provide informed consent
* Students and/or parents who do not provide a telephone number and e-mail address to be contacted

Ages: 11 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Children's vaccination uptake | 90 days
  Measured through a telephonic interview to parents, difference in vaccination rates (% before/after)
Children's knowledge on HPV vaccination | 90
  Measured through: (1) the Questionnaire - HAVIQ Adolescente Vaccine Intervention Questionnaire; 5-point Likert scale (from 1=strongly disagree to 5=strongly agree). (2) 10 items with dichotomous "yes/no" responses. Each correct answer will be assigned a score of 1, each answer not given or incorrect, zero. The total score ranges from 0 (no knowledge) to 10 (highest level of knowledge).
Children's self-efficacy in receiving the vaccine | 90
  Measured through the Questionnaire - HAVIQ Adolescente Vaccine Intervention Questionnaire; 100-point scale (0="not at all confident"; 100="completely confident").
Children's fear and anxiety towards vaccination | 90
  Measured through the Questionnaire - HAVIQ Adolescente Vaccine Intervention Questionnaire; 5-point Likert scale (from 1=strongly disagree to 5=strongly agree)
Children's involvement in vaccine decision making | 90
  Measured through the Questionnaire - HAVIQ Adolescente Vaccine Intervention Questionnaire; 5-point Likert scale (from 1=strongly disagree to 5=strongly agree)

SECONDARY OUTCOMES:
Parent's hesitancy about vaccination | 90 days
  Measured through the Questionnaire - Parent Attitudes about Childhood Vaccines Survey (PACV) - The total score ranges from 0 to 100: a parent is considered non-hesitant if he or she scores <50 and hesitant with a value of ≥50

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Cicolini, Principal Investigator — Researcher
Locations (1):
- University Aldo Moro of Bari, Bari, Apulia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Napolitano F, D'Alessandro A, Angelillo IF. Investigating Italian parents' vaccine hesitancy: A cross-sectional survey. Hum Vaccin Immunother. 2018 Jul 3;14(7):1558-1565. doi: 10.1080/21645515.2018.1463943. Epub 2018 May 14. PMID 29641945
- [Background] Forster AS, McBride KA, Davies C, Stoney T, Marshall H, McGeechan K, Cooper SC, Skinner SR. Development and validation of measures to evaluate adolescents' knowledge about human papillomavirus (HPV), involvement in HPV vaccine decision-making, self-efficacy to receive the vaccine and fear and anxiety. Public Health. 2017 Jun;147:77-83. doi: 10.1016/j.puhe.2017.02.006. Epub 2017 Mar 18. PMID 28404501
- [Background] Opel DJ, Taylor JA, Mangione-Smith R, Solomon C, Zhao C, Catz S, Martin D. Validity and reliability of a survey to identify vaccine-hesitant parents. Vaccine. 2011 Sep 2;29(38):6598-605. doi: 10.1016/j.vaccine.2011.06.115. Epub 2011 Jul 16. PMID 21763384
- [Background] Gottvall M, Tyden T, Hoglund AT, Larsson M. Knowledge of human papillomavirus among high school students can be increased by an educational intervention. Int J STD AIDS. 2010 Aug;21(8):558-62. doi: 10.1258/ijsa.2010.010063. PMID 20975088